CLINICAL TRIAL: NCT04643275
Title: Effect of BTL-899 Device for Non-invasive Lipolysis on Human Upper Arms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-899A
Record Dates: First submitted 2020-11-03; First posted 2020-11-25 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Fat Burn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Non-invasive lipolysis of the upper arms (Experimental): The treatment administration phase consists of four (4) treatment visits, delivered 5- 10 - days apart. Each therapy session will last 30 minutes. Follow-ups visits at 1 month and 3 months after the final treatment will be held.
  Interventions: Device: BTL-899

INTERVENTIONS:
Device: BTL-899 — Treatment with study device.

SUMMARY:
This study will evaluate the clinical safety and the performance of the BTL-899 device during the treatment of upper arms.

DETAILED DESCRIPTION:
The aim of the study is to confirm the efficacy and the safety of the treatment. The efficacy (reduction of excess adipose tissue) will be assessed via correct identification of pre-treatment and 3-months follow-up images by at least two out of three independent blinded evaluators. The fat reduction will be also measured by means of ultrasound. Comfort and satisfaction will be assessed via standard questionnaires.

Safety measures will include documentation of adverse events (AE) during and after the procedures.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 20 to 35 kg/m2.
* Visible excess of adipose tissue at the treatment site
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring and/or weight loss during study participation.
* No procedure for fat reduction in the area in the last six months.
* Subjects willing and able to maintain his/her regular (pre-procedure) diet and exercise regimen without effecting a significant change of weight in either direction during the study participation.

Exclusion Criteria:

* Electronic implants (such as cardiac pacemakers, defibrillators, and neurostimulators)
* Cardiovascular diseases
* Vascular diseases (such as chronic venous insufficiency, deep venous thrombosis, varicose veins, etc.)
* Disturbance of temperature or pain perception
* Pulmonary insufficiency
* Metal implants
* Drug pumps
* Malignant tumor
* Hemorrhagic conditions
* Septic conditions and empyema
* Acute inflammations
* Systemic or local infection such as osteomyelitis and tuberculosis
* Contagious skin disease
* Elevated body temperature
* Pregnancy
* Breastfeeding
* Injured or otherwise impaired muscles in the arms
* Scars, open lesions, and wounds at the treatment area
* Basedow's disease
* Previous liposuction in the treatment area in the last six months
* Any other disease or condition at the investigator's discretion, e.g. dislocated shoulder or carpal tunnel syndrome than can pose danger to the patient or compromise the study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Statistically significant reduction of fat thickness in the upper arms evaluated by photographs | 5 months
  To gather clinical evidence that the BTL-899 device is able to induce non-invasive lipolysis when used on upper arms. The primary efficacy outcome measure is a minimum 75% of the subjects' pre-treatment and 3-months follow-up images to be correctly identified by at least two of three independent blinded evaluators.

SECONDARY OUTCOMES:
Evaluation of the Therapy's Safety Measured Via Therapy Comfort Questionnaire | 7 months
  Assessment the safety of the BTL-899 device when used for non-invasive lipolysis of the upper arms via questionnaires filled in by the participants following each therapy session. On Numerical Analog Scale (0-10), where 0 represents 'no pain' and 10 represents 'worst possible pain' select the level of pain experienced during the treatment. The outcome will further be measured through the occurrence of adverse events or lack thereof.
Evaluation of the participants' satisfaction with the therapy evaluated via standard questionnaires | 5 months
  Evaluation of the participants' satisfaction with the therapy and the results. ● Minimum 80% of treated subjects to report satisfaction (level satisfied and higher) with the therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Denkova Dermatology, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No